CLINICAL TRIAL: NCT04195087
Title: Perfusion Index and Pleth Variability Index in Predicting Hypotension Following Spinal Anesthesia Performed in Sitting Position in Cesarean Section.
Brief Title: Perfusion Index and Pleth Variability Index in Cesarean Section.
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Ozyurt, Study director, Antalya Training and Research Hospital
Other Study IDs: AntalyaEAH02
Record Dates: First submitted 2019-12-02; First posted 2019-12-11 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; perfusion index; Pleth variability index; sitting position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-hypotension: Patients with a mean arterial pressure reduction of less than 20% and/or systolic arterial pressure above 80 mmHg after spinal anesthesia.
  Interventions: Device: Masimo Radical-7® Pulse CO-Oximeter®
- Hypotension: Patients with a 20% reduction in mean arterial pressure and/or systolic arterial pressure below 80 mmHg after spinal anesthesia.
  Interventions: Device: Masimo Radical-7® Pulse CO-Oximeter®

INTERVENTIONS:
Device: Masimo Radical-7® Pulse CO-Oximeter® — The perfusion index and Pleth variability index will be recorded from the device monitor.

SUMMARY:
The aim of this study is to investigate the predictability of hypotension by using PI and PVI in pre-and post-spinal anesthesia periods in cesarean section cases in the sitting position.

DETAILED DESCRIPTION:
Spinal anesthesia has been widely used all over the world due to its superiority to general anesthesia in cesarean section. However, as a result of the sympathetic blockade in spinal anesthesia, vascular tone decreases and hypotension occurs. The incidence of hypotension increases up to 70% in pregnant women due to increased sensitivity to local anesthetics and increased intraabdominal pressure. Improper management of postspinal hypotension may lead to maternal and fetal complications. Predicting the risk of hypotension in patients undergoing spinal anesthesia may allow applications such as volume loading or prophylactic vasopressor use. The perfusion index, measured by pulse Oximeters, correlates with blood flow changes at the tip of the finger so that it can detect hypotension and thus decrease in blood flow after spinal anesthesia. Pleth variability index (PVI) is a non-invasive value found in the new generation pulse oximeters. It is a parameter used in the dynamic measurement of response to fluid therapy in intensive care units. PVI can dynamically give an idea about the fluid status of the pregnant woman. Previous studies have shown that PVI may be a marker for predicting hypotension following spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who will undergo elective cesarean section

Exclusion Criteria:

* Preeclampsia
* Cardiovascular disorder
* Fetal abnormality
* Patients who failed spinal anesthesia or switched to general anesthesia during operation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who will undergo elective cesarean section
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Perfusion index | Before spinal anesthesia in supine positon
  Perfusion index will be recorded from the monitor.
Pleth variability index | Before spinal anesthesia in supine positon
  Pleth variability index will be recorded from the monitor.
Perfusion index | Before spinal anesthesia in sitting positon
  Perfusion index will be recorded from the monitor.
Pleth variability index | Before spinal anesthesia in sitting positon
  Pleth variability index will be recorded from the monitor.
Perfusion index | 1 minutes after spinal anesthesia in supine positon
  Perfusion index will be recorded from the monitor.
Pleth variability index | 1 minutes after spinal anesthesia in supine positon
  Pleth variability index will be recorded from the monitor.
Perfusion index | Start of the surgery
  Perfusion index will be recorded from the monitor.
Pleth variability index | Start of the surgery
  Pleth variability index will be recorded from the monitor.
Perfusion index | 1 minutes after the umbilical cord clamping
  Perfusion index will be recorded from the monitor.
Pleth variability index | 1 minutes after the umbilical cord clamping
  Pleth variability index will be recorded from the monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan OZYURT, MD, Study Director — University of Health Sciences, Antalya Training and Research Hospital
Locations (1):
- University of Health Sciences, Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)